CLINICAL TRIAL: NCT04302324
Title: A Phase II Study of Daratumumab, Clarithromycin, Pomalidomide And Dexamethasone (D-ClaPd) In Multiple Myeloma Patients Previously Exposed to Daratumumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-12021155
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma; Relapse Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- daratumumab/clarithromycin/pomalidomide/dexamethasone (Experimental): Induction Phase: 8 cycles (cycle length of 28 days)
  * Daratumumab SC:
    1800mg SC weekly for 8 weeks for Cycle 1 and 2 1800mg SC every 2 weeks on Day 1 and 15 for Cycle 3-6 1800mg SC every 4 weeks on Day 1 for Cycle 7-8
  * Clarithromycin
    500mg PO BID until VGPR or 8 cycles, whichever occurs first
  * Pomalidomide 4mg PO on Days 1-21
  * Dexamethasone 20mg IV as pre-medication on Day 1, 8 40mg PO on the day after daratumumab for Cycle 1 Days 15 and 22 40mg PO pre-daratumumab weekly for Cycle 2-6 20mg PO pre-daratumumab weekly for Cycle 7-8
  Maintenance Phase (Cycle 9+): Up to 24 cycles (cycle length of 28 days)
  * Daratumumab 1800 mg SC on Day 1
  * Pomalidomide 4mg PO on Day 1-21
  * Dexamethasone 20mg PO pre-daratumumab weekly for Cycles 9 and beyond
  Interventions: Drug: Daratumumab SC; Drug: Clarithromycin; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab SC — Given as 1800mg via injection
  Other Names: Faspro
Drug: Clarithromycin — Given as 500mg oral capsule
Drug: Pomalidomide — Given as 4mg oral capsule
Drug: Dexamethasone — Given as 20mg IV and 20mg or 40mg oral tablets

SUMMARY:
This is a single-center, non-randomized, phase 2 study in which patients will receive daratumumab (subcutaneous, SC) in combination with clarithromycin/pomalidomide/dexamethasone (D-ClaPd) until progressive disease (PD) or unacceptable toxicity. This study will test the hypothesis that in patients with previous daratumumab exposure, combination therapy of clarithromycin/pomalidomide/dexamethasone with daratumumab SC (D-ClaPd) will yield higher Very Good Partial Response (VGPR) rates in relapsed/refractory multiple myeloma patients than historical pomalidomide/dexamethasone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Multiple Myeloma
* Relapsed and/or refractory myeloma defined as follows: Relapse or progressive disease after at least one previous line of therapy which must include prior daratumumab. At least 8 doses of daratumumab in a previous line must be administered either as monotherapy or in combination with a daratumumab-free interval of ≥3 months AND patient may be daratumumab refractory defined as less than a partial remission (PR) achieved on prior daratumumab-based therapy or have exhibited progression within 60 days of receiving daratumumab. If previous therapy was autologous stem cell transplant (SCT), over 3 months must have elapsed after SCT.
* Measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >0.1 g/dL serum free light chains, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* Females of childbearing potential(FCBP) must have a negative serum or urine pregnancy test within 10 - 14 days prior to and again within 24 hours of prescribing pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Able to take aspirin daily
* Life expectancy must be greater than 3 months.
* Be able to voluntarily sign and understand written informed consent.
* Absolute neutrophil count (ANC) ≥750 cells/mm3 (.75 x 109/L)
* Platelets count ≥ 50,000/mm3 (50 x 109/L)
* Serum SGOT/AST ≤ 2.0 x upper limits of normal
* Serum SGPT/ALT <3.0 x upper limits of normal
* Serum creatinine ≤ 2.5 x upper limits of normal
* Serum total bilirubin ≤ 1.5 x upper limits of normal (Total bilirubin ≥ 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* All participants must be registered into the mandatory POMALYST REMS™ program and be willing and able to comply with the requirements of the POMALYST REMS™ program.

Exclusion Criteria:

* Prior exposure to non-daratumumab anti-CD38 monoclonal antibodies or pomalidomide. Prior pomalidomide exposure in 1 or more previous lines of therapy allowed if partial remission (PR) or better achieved. No disease progression may have occurred within 60 days of receiving pomalidomide.
* New York Heart Association (NYHA) Class III or IV heart failure, unstable cardiac arrhythmia, or unstable angina
* Myocardial infarction within the past 6 months
* Severe obstructive airway disease
* Planned high-dose chemotherapy and autologous stem cell transplantation within 6, 28-day treatment cycles after starting on treatment
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment (if area involved is small than within 7 days)
* Systemic treatment, within 14 days before the first dose, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Seropositive for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has greater than Grade 3 peripheral neuropathy, or Grade 2 pain
* Participation in other clinical trials within 30 days
* History of thromboembolic event within the past 6 months prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Very Good Partial Response Rate or better within 8 cycles of induction therapy | 8 months
  Very Good Partial Response or better defined as the proportion of participants with a documented Very Good Partial Response (VGPR) or better as best response per International Myeloma Working Group (IMWG) criteria, measured from date of enrollment through the end of the 8th induction cycle.

SECONDARY OUTCOMES:
Progression-Free Survival | Approximately 3 years
  Progression-Free Survival (PFS) is measured in months from the date of enrollment to the date of disease progression and/or death. Median estimate is calculated using the Kaplan-Meier methodology.
Overall Survival | Approximately 5 years
  Overall Survival (OS) is measured in months from the date of enrollment to the date of the participant's death. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier survival estimates.
Complete Response Rate or Better | Approximately 1 year
  The proportion of participants with a documented Complete Response (CR) or better, per International Myeloma Working Group (IMWG) criteria.
Time to Progression | Approximately 3 years
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met the criteria for Progressive Disease
Time to Next Therapy | Approximately 3 years
  Measured in months from the date of enrollment to the start date of subsequent treatment for relapsed/refractory multiple myeloma
Duration of Response | Approximately 3 years
  Duration of Response (DoR) is defined as the time between the date of initial documentation of best response to the date of first documented evidence of disease progression.
Rate of minimal residual disease (MRD) negativity | Approximately 8 months
  Defined as a percentage of MRD negative participants
Rate of improvement in response during maintenance therapy | Approximately 3 years
  Percentage of patients that achieved an improved response during maintenance compared to end of induction.
Time to Best Response | Approximately 8 months
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met criteria for best response per International Myeloma Working Group (IMWG) criteria.
Overall Response Rate | Approximately 1 year
  The proportion of participants with a documented Overall Response (Partial Response or better), per International Myeloma Working Group (IMWG) criteria.
Very Good Partial Response (VGPR) Rate or better | Approximately 1 year
  The proportion of participants with a documented Very Good Partial Response (VGPR) Rate or better, per International Myeloma Working Group (IMWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Rosenbaum, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine - Multiple Myeloma Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No